CLINICAL TRIAL: NCT00002751
Title: PROTOCOL FOR A PHASE I STUDY OF INTRATHECAL MONOCLONAL ANTIBODY FRAGMENT 131I Me1-14 F(ab')2 IN PATIENTS WITH NEOPLASMS METASTATIC TO THE LEPTOMENINGES
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Brain Metastases
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Darell Bigner, MD, Duke UMC
Purpose: Treatment
Other Study IDs: 1193; DUMC-1193-006R11; DUMC-1017-96-7R7; DUMC-1100-97-7R8; DUMC-1159-98-7R9; DUMC-1229-99-7R10; DUMC-657897; DUMC-997-95-7R6; NCI-V90-0052; NCI-H96-0010; CDR0000064687 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-07-01 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2009-10

CONDITIONS: Metastatic Cancer
Keywords: leptomeningeal metastases
MeSH Terms: conditions — Neoplasm Metastasis; Meningeal Carcinomatosis

INTERVENTIONS:
Biological: monoclonal antibody Me1-14 F(ab')2

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody therapy in treating patients who have brain metastases.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicity and maximum tolerated dose of 131-iodine-labeled monoclonal antibody fragment Me1-14 F(ab')2 administered intrathecally in patients with neoplasms metastatic to the leptomeninges. II. Identify objective therapeutic responses to this treatment.

OUTLINE: Radioimmunotherapy. Iodine-131-Labeled Monoclonal Antibody Fragment Me1-14 F(ab')2, 131I-Me1-14 F(ab')2.

PROJECTED ACCRUAL: Three to 6 patients will be treated at each dose studied.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed neoplasm that is recurrent in the subarachnoid space Biopsy of recurrent lesion required if original diagnosis made more than 2 years prior to entry and CSF cytology negative Radiographic evidence of measurable lesion in the leptomeninges (by myelography, CT, or MRI) or cytologic evidence of malignancy in the CSF Any type of neoplasm eligible provided tumor cells (tissue or CSF preparation) bind significantly to intact monoclonal antibody Me1-14 IgG2a or to Me1-14 F(ab')2 Patency of subarachnoid pathways demonstrated by isotopic intraventricular flow

PATIENT CHARACTERISTICS: Age: 3 and over Performance status: Karnofsky 50-100% Hematopoietic: Absolute neutrophil count at least 1,000/mm3 Platelet count at least 100,000/mm3 Hepatic: AST less than 1.5 times upper limit of normal (ULN) Alkaline phosphatase less than 1.5 times ULN Renal: Creatinine less than 1.2 mg/dL Other: No allergy to iodine Not pregnant or nursing

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior antineoplastic chemotherapy unless unequivocal evidence of tumor progression No concurrent systemic chemotherapy Endocrine therapy: Corticosteroids allowed if at lowest possible dose and stable for at least 10 days prior to entry Radiotherapy: At least 3 months since prior radiotherapy to site of measurable disease unless unequivocal evidence of disease progression Surgery: Not specified

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 1989-07; Study Completion 2004-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darell D. Bigner, MD, PhD, Study Chair — Duke University
Locations (1):
- Duke Comprehensive Cancer Center, Durham, North Carolina, United States